CLINICAL TRIAL: NCT04637334
Title: Superior Vena Cava Reconstruction in Patients on Hemodialysis
Acronym: Hemodialysis
Status: Completed | Type: Observational
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 2013.00.642.A
Record Dates: First submitted 2019-08-12; First posted 2020-11-19 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Superior Vena Cava Syndrome
MeSH Terms: conditions — Superior Vena Cava Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Superior vena cava reconstruction — Endovascular therapy with percutaneous transluminal angioplasty (PTA) and, in recent years, with stenting of the SVC, has been performed with increasing frequency. An endovascular approach is the current standard of care to relieve SVC obstruction due to malignancy to obtain prompt relief of the rapidly emerging symptoms and improve quality of life,3 keeping in mind the short life expectancy of these patients. The role of endovascular therapy in SVC syndrome of nonmalignant etiology is undecided because long-term durability of this treatment method remains to be assessed.

SUMMARY:
The treatment objective for patients with SVC syndrome secondary to both malignant and benign etiologies is to reduce the elevated central venous pressures.1 However, the strategies are contingent upon the underlying disease process. Thus the management of SVC syndrome ranges from medical or supportive care to surgical bypass,3 and it is important for physicians to understand the varied treatment modalities of this potentially life-threatening disease.17 Fortunately, the overwhelming majority of patients with SVC syndrome secondary to benign causes develop a physiologic compensation for the obstruction that can be treated with anticoagulation and endovascular modalities. Intervention for symptomatic relief may not be required.1 An endovascular approach is the current standard of care to relieve SVC obstruction due to malignancy to obtain prompt relief of the rapidly emerging symptoms and improve quality of life,3 keeping in mind the short life expectancy of these patients. The role of endovascular therapy in SVC syndrome of nonmalignant etiology is undecided because the long-term durability of this treatment method remains to be assessed.

DETAILED DESCRIPTION:
This case study will retrospectively review all SVC syndrome and/or occlusion procedures since January 2009. All patients were given adequate informed consent about the procedure and its benefits and complications.

Definitions of clinical outcomes will adhere to the Subcommittee on Reporting Standards in Venous disease.27 Risk factors and outcomes of these procedures will be retrospectively analyzed. Data collected included preoperative patient demographics, clinical status, noninvasive and invasive imaging, operative procedural details, post-operative complications, post-procedural imaging surveillance, adjunctive/re-intervention procedures, clinical outcome during follow-up, and mortality. Primary endpoints will be clinical outcome and patency. Secondary endpoints will be re-intervention rate and death within 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Presence of SVC syndrome or SVC occlusion
* Presence of ESRD on hemodialysis
* Presence of upper extremity or neck access, either catheter or surgical fistula
* Patients who have received endovenous or open bypass reconstruction of the SVC secondary to SVC syndrome or SVC occlusion

Exclusion Criteria:

* Patients who have not undergone endovenous or open bypass reconstruction of the SVC secondary to SVC syndrome or SVC occlusion

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who underwent SVC bypass procedures from January 2010 to June 2013 at Methodist Dallas Medical Center will be screened for participation in the study.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2014-09-13 (Actual); Primary Completion 2022-05-06 (Actual); Study Completion 2022-05-06 (Actual)

PRIMARY OUTCOMES:
Clinical outcome and patency | Upto 30 days
  To report findings in patients with ESRD on hemodialysis who underwent SVC reconstruction

CONTACTS AND LOCATIONS:
Overall Officials: Robert Feldtman, M.D., Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided